CLINICAL TRIAL: NCT00340574
Title: Phase I Study of the Safety and Immunogenicity of AMA-1-C1/Alhydrogel + CPG 7909, An Asexual Blood Stage Vaccine for Plasmodium Falciparum Malaria
Brief Title: Improving the Efficacy of Experimental Malaria Vaccine AMA1-C1/Alhydrogel® (Registered Trademark)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905117; 05-I-N117
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-02

CONDITIONS: Healthy Volunteer; HV
Keywords: Human; Clinical Trial; Mosquito; Healthy Volunteer; HV
MeSH Terms: interventions — ProMune

INTERVENTIONS:
Drug: AMA1-C1/Alhydrogel + CpG 7909

SUMMARY:
This study will evaluate the safety and efficacy of the experimental malaria vaccine AMA1-C1/Alhydrogel® (Registered Trademark) and determine whether a new, additional component of the vaccine may increase its effectiveness. Malaria is a debilitating and potentially fatal blood disease transmitted by a parasite found in certain mosquitoes. The AMA1-C1 vaccine has been designed to create an immune response against the parasite and prevent the disease. The purpose of the study is to determine whether the additional component-protein pieces known as CpG- improves the immune response to the vaccine without causing problematic side effects.

Volunteers must be healthy adults between 18 and 45 years old. Individuals who have had malaria in the past or have recently traveled to areas where malaria is endemic will be excluded from the study. Candidates will be screened with a physical examination, blood tests, and medical history.

Participants will be involved in a three-stage study. In the first stage, a group of participants will receive either a high dose of the vaccine alone or a low dose combined with the CpG protein. In the second stage, a different group of participants will receive a high dose of the vaccine alone or a high dose combined with CpG. In the third stage, a larger group of participants will receive a high dose of the vaccine alone or a high dose combined with CpG. The vaccine will be injected into the muscle of the upper arm, and all participants will receive three doses of the vaccine with 28 days between doses to monitor possible reactions and side effects. Participants will be monitored for 30 minutes after each injection and will record any symptoms they experience over the six days after receiving their dose. In addition, participants will be examined over the course of six months during and after the trial with physical exams and blood and urine tests.

DETAILED DESCRIPTION:
Purpose: This study will evaluate the safety and immunogenicity of the experimental malaria vaccine AMA1-C1/Alhydrogel® (Registered Trademark), and the ability of the TLR-9 agonist CPG 7909 oligodexoynucleotide (ODN) to augment antibody response to the vaccine and alter the Th1/Th2 bias. The vaccine preparations to be studied contain an equal mixture of AMA1 from two different clones of Plasmodium falciparum (FVO and 3D7), both produced separately as recombinant proteins expressed by Pichia pastoris (PpAMA-1 FVO and PpAMA-1 3D7). Bulk PpAMA-1 antigens were purified from culture medium of transformed yeast grown in a 60L fermenter. The correctly folded PpAMA-1 was purified from this mixture by a combination of affinity, ionic, hydrophobic and gel filtration chromatography. Purified PpAMA-1 FVO and PpAMA-1 3D7 were subsequently mixed and adsorbed onto aluminum hydroxide gel (Alhydrogel® (Registered Trademark)). The CPG 7909 ODN formulation used in this study (CPG 7909) is manufactured by Coley Pharmaceutical Group. Subjects will be randomly assigned to receive Alhydrogel® (Registered Trademark) formulated vaccine with or without CPG 7909 in a point of use formulation.

Research Environment: The study will be conducted at the University of Rochester Vaccine and Treatment Evaluation Unit (VTEU).

Subjects: Subjects for this study will be healthy adults between the ages of 18 and 45 years with no history of malaria or of recent travel to malaria-endemic areas. Subjects will be enrolled in three consecutive dose-escalation cohorts with review by a Safety Monitoring Committee between cohorts.

Subject participation: Subjects will receive three vaccinations with the AMA1-C1/Alhydrogel® (Registered Trademark) vaccine formulated in Alhydrogel® (Registered Trademark) with or without CPG 7909 adjuvant over 2 months (0, 1, 2 months) by intramuscular (IM) injection. Subjects will have multiple blood samples obtained over the next 6 months.

Variables to be Investigated: Samples will be tested for binding antibody to AMA1 and for ability to inhibit the growth of plasmodia in vitro. In addition, antigen-specific activated B cells in peripheral blood will be enumerated, as well as the relative ratio of antigen-specific Th1-like and Th2-like T cells.

Risk/Benefits: The risks of participating in this study are those associated with administration of AMA1-C1/Alhydrogel® (Registered Trademark) and of CPG 7909, and include local pain, systemic inflammatory responses including fever and influenza-like symptoms, and induction of autoimmune responses. As with any other investigational vaccine, there are unknown risks. Subjects may derive no benefit from participation in this study. Development of effective vaccines to prevent malaria is an important societal benefit.

Confidentiality: Volunteers will have code numbers and will not be identified by name.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age between 18 and 45 years, inclusive.

Good general health as a result of review of medical history and/or clinical tests.

Available for the duration of the trial (34 weeks).

Willingness to participate in the study as evidenced by signing the informed consent document.

EXCLUSION CRITERIA:

Pregnancy as determined by a positive urine beta-hCG (if female) at any point during the study.

Participant unwilling to use highly effective contraception methods (such as: abstinence, birth control pills or birth control patches or vaginal ring, diaphragm with spermicide, IUD (intrauterine device), condom with spermicide, progestin implant or injection, surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation), or a partner who has had a vasectomy for the duration of the trial (if female).

Currently lactating and breast-feeding (if female).

Evidence of clinically significant immunosuppressive, neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.

Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the volunteer to understand and cooperate with the study protocol.

Laboratory evidence of liver disease (aspartate aminotransferase greater than 1.25 times the upper limit of normal of the testing laboratory).

Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory).

Laboratory evidence of hematologic disease (absolute neutrophil count less than 1,500/mm3; hemoglobin less than 0.9 times the lower limit of normal of the testing laboratory, by sex; or platelet count less than 140,000/mm3).

Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

Participation in another investigational vaccine or drug trial within the 30 days of starting this study or while this study is ongoing.

Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.

History of a severe allergic reaction or anaphylaxis.

Severe asthma (emergency room visit or hospitalization within the last 6 months).

Serologic evidence of infection with HIV-1, HBV, or HCV.

Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or while the study is ongoing.

Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.

History of a surgical splenectomy.

Receipt of blood products within the past 6 months.

Previous receipt of an investigational malaria vaccine.

Receipt of antimalarial prophylaxis during the past 12 months.

Prior malaria infection.

Travel to a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.

History of a known allergy to nickel.

Pre-existing autoimmune or antibody mediated diseases including but not limited to: systemic lupus erythematosis, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia; or laboratory evidence of possible autoimmune disease determined by a positive anti-dsDNA titer, positive rheumatoid factor, proteinuria and/or a positive ANA.

Chloroquine and related compounds within 12 weeks of study entry.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 2005-03-08; Study Completion 2008-07-02

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - National Institute of Allergy and Infectious Diseases (NIAID), 9000 Rockville Pi, Bethesda, Maryland
  - University of Rochester, Rochester, New York

REFERENCES:
- [Background] Waters AP, Thomas AW, Deans JA, Mitchell GH, Hudson DE, Miller LH, McCutchan TF, Cohen S. A merozoite receptor protein from Plasmodium knowlesi is highly conserved and distributed throughout Plasmodium. J Biol Chem. 1990 Oct 15;265(29):17974-9. PMID 2211675